CLINICAL TRIAL: NCT00521794
Title: Andersen-Tawil Syndrome: Genotype-Phenotype Correlation and Longitudinal Study
Brief Title: Characteristics of Andersen-Tawil Syndrome
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Robert Griggs, MD, Professor of Neurology, Medicine, Pediatrics, Pathology & Laboratory Medicine, and Center for Human Experimental Therapeutics, University of Rochester
Other Study IDs: RDCRN 5301; 5U54RR019482-02 (NIH)
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Andersen-Tawil Syndrome; Andersen Syndrome
Keywords: Arrhythmia; Muscle Weakness; Periodic Paralysis; Channelopathy
MeSH Terms: conditions — Andersen Syndrome; Arrhythmias, Cardiac; Muscle Weakness; Channelopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Andersen-Tawil Syndrome (ATS) is a rare, genetic disorder that causes episodes of muscle weakness, potentially life-threatening changes in heart rhythm, and developmental abnormalities. Disease symptoms can vary, the cause of some ATS cases remains unknown, and no specific treatment has been identified. The purpose of this multi-site study is to better characterize ATS, establish whether symptoms change over time, and determine if symptoms are related to a mutation in the KCNJ2 gene.

DETAILED DESCRIPTION:
ATS is an ion channel disorder that causes episodes of muscle weakness and potentially life-threatening heart arrhythmias for which no treatment has been identified. The majority of ATS cases are caused by a mutation in the KCNJ2 gene; other cases result from unknown causes. The KCNJ2 gene mutation alters potassium channels in such a way that it disrupts the flow of potassium ions in skeletal and heart muscle. This can lead to the characteristic periodic paralysis and irregular heart rhythms. The purpose of this study is to better define the genetic basis, clinical features, and disease progression of ATS. The study will also establish clinically relevant endpoints for use in future clinical studies.

This observational study will last 2 years and will involve three study visits. The first visit will entail a 1.5- to 3.5-day inpatient stay; the length of stay will depend on whether a participant has been taking medications for their symptoms of weakness. Participants will be asked to discontinue use of such medications during the inpatient stay. Participants will not be asked to stop any medications that they may be taking for heart symptoms. This first study visit will include a medical history, a quality of life questionnaire, a physical exam, and muscle strength testing. Nerve, muscle, and heart activity will also be measured, and blood will be drawn for laboratory tests and optional DNA analysis. The second and third study visits will take place 1 and 2 years after the initial study visit and will include the same evaluations. During the 8 weeks following each study visit, participants will record in a telephone diary any muscle and heart symptoms that they experience. During the 1 week after both yearly visits, participants will also undergo an outpatient heart rhythm evaluation. A study coordinator will contact participants once a month by phone over the course of the study to review symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of ATS as defined by at least two of the following three criteria:

  1. Presence of clear-cut episodes of transient muscle weakness with or without a fixed deficit, typically following exertion or prolonged rest OR atypical history with otherwise typical exam findings (absent reflexes with normal sensation during an episode) OR unexplained hypokalemia between episodes OR abnormal long-exercise nerve conduction study
  2. Heart conduction defects: prolonged QTc interval on 12-lead electrocardiogram OR ventricular ectopy, including uniform or multifocal PVCs, polymorphic VT, or bidirectional VT
  3. Presence of two or more of the following physical features: low set ears, hypertelorism, small mandible, clinodactyly, syndactyly, micromelia of hands or feet --OR--
* Meets one of the above three criteria and has at least one family member with two of the criteria --OR--
* Does not meet the above three criteria, but possesses a mutation in the KCNJ2 gene

Exclusion Criteria:

* Less than 10 years of age

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a clinically confirmed diagnosis of Andersen-Tawil Syndrome (ATS) enrolled across seven sites in the United States, England, Italy and Canada
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Collect prospective standardized data from participants to help better define the clinical phenotype of ATS. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emma Ciafaloni, MD, Study Chair — University of Rochester; Robert C. Griggs, MD, Principal Investigator — University of Rochester
Locations (7):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Rochester School of Medicine and Dentistry, Rochester, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- London Health Sciences Centre, London, Ontario, Canada
- University of Milan, Milan, Italy
- Institute of Neurology and National Hospital for Neurology, London, United Kingdom

REFERENCES:
- [Background] Tawil R, Ptacek LJ, Pavlakis SG, DeVivo DC, Penn AS, Ozdemir C, Griggs RC. Andersen's syndrome: potassium-sensitive periodic paralysis, ventricular ectopy, and dysmorphic features. Ann Neurol. 1994 Mar;35(3):326-30. doi: 10.1002/ana.410350313. PMID 8080508
- [Background] Sansone V, Griggs RC, Meola G, Ptacek LJ, Barohn R, Iannaccone S, Bryan W, Baker N, Janas SJ, Scott W, Ririe D, Tawil R. Andersen's syndrome: a distinct periodic paralysis. Ann Neurol. 1997 Sep;42(3):305-12. doi: 10.1002/ana.410420306. PMID 9307251
- [Background] Tristani-Firouzi M, Jensen JL, Donaldson MR, Sansone V, Meola G, Hahn A, Bendahhou S, Kwiecinski H, Fidzianska A, Plaster N, Fu YH, Ptacek LJ, Tawil R. Functional and clinical characterization of KCNJ2 mutations associated with LQT7 (Andersen syndrome). J Clin Invest. 2002 Aug;110(3):381-8. doi: 10.1172/JCI15183. PMID 12163457